CLINICAL TRIAL: NCT06196931
Title: Clinical Value of DWI-ADC Matching in the Short-term Prognosis of Wilson's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Affiliated to the Institute of Neurology, Anhui University of Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: AHnkyy20231020
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Hepatolenticular Degeneration; Wilson
Keywords: DWI-ADC matching; Wilson disease; clinical value; short-term prognosis
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In earlier studies, it was found that patients of Wilson disease with new diagnosed who only has neurological symptoms often had DWI hyper-intensity in brain MRI, which was more common in putamen and midbrain, indicating that the disease was in the acute stage. However, many patients had ADC hyper-intensity or hypo-intensity at the same time, and the two different signals represented different disease processes from an imaging perspective. The former indicating T2 penetration effect, and the latter represents diffusion limitation, which indicating the presence of local inflammation, edema, etc. Whether the signal changes of these two different matching modes have guiding significance for the early de-copper treatment for WD, one is the core point of our study. We hope to exploring the predictive value about DWI-ACD signal matching for symptoms changes in the earlier time of de-copper treatment through this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients had been previously diagnosed with WD who both had DWI hyper-intensity and ADC hyper-intensity or hypo-intensity at the same time；
2. Patients who accept de-copper treatment in hospitalization for 4 weeks or more.

   Exclusion Criteria:
   1. Patients who only with liver injury;
   2. Severe complications;
3. Combined with other diseases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: WD should be considered in patients with unexplained liver disease, neurological symptoms (especially extrapyramidal symptoms), or psychiatric symptoms. Age of onset cannot be used as a basis for diagnosing or ruling out WD.
  Among these, patients had been previously diagnosed with WD who both had DWI hyper-intensity and ADC hyper-intensity or hypo-intensity at the same time. At the time of admission, the Unified Wilson Disease Rating Scale (UWDRS) and cranial MRI examinations were conducted to assess the state of the disease. All patients received Cu-chelating therapy according to the Chinese guidelines for the diagnosis and treatment of WD (Neurogenetics Group and Neurology Branch of Chinese Medical Association, 2021). During the course of treatment, serum copper, ceruloplasmin, and urine copper at 24 h before treatment and the highest urine copper at 24 h during treatment were tested to determine the efficacy of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
UWDRS scales | Before and 4 weeks after treatment
  It is used to evaluate the changes of patients' nervous system symptoms
24h urine copper | Before and 4 weeks after treatment
  used to evaluate the changes of patients' nervous system symptoms

SECONDARY OUTCOMES:
Semi-quantitative brain MRI score | Before de-copper treatment
  It is used to evaluate the changes of patients' nervous system symptoms
ALT, AST and other liver function test | Before and 4 weeks after treatment
  used to evaluate the changes of patients' nervous system symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- The affiliated hospital of Institute of Neurology in Anhui University of Chinese Medicine, Hefei, Anhui, China